CLINICAL TRIAL: NCT04648891
Title: Spasmodic Dysphonia Pain Study
Brief Title: Spasmodic Dysphonia Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David G. Lott, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-006889
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Spasmodic Dysphonia
Keywords: Pain
MeSH Terms: conditions — Dysphonia; Pain | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients will receive standard of care laryngeal injection of Botox via a transcricothyroid approach without additional anesthesia
- Lidocaine (Experimental): Patients will receive standard of care laryngeal injection of Botox via a transcricothyroid approach following subcutaneous injection of lidocaine (approximately 2 minutes before Botox injection).
  Interventions: Drug: Lidocaine
- Vibrating Wand (Experimental): Patients will receive standard of care laryngeal injection of Botox via a transcricothyroid approach while using the vibrating wand.
  Interventions: Device: Vibrating wand

INTERVENTIONS:
Drug: Lidocaine — Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
  Arms: Lidocaine
Device: Vibrating wand — a vibrating instrument held adjacent to the cricothyroid space
  Arms: Vibrating Wand

SUMMARY:
This study aims to identify adjuvant methods to improve patient comfort during in-office laryngology procedures.

DETAILED DESCRIPTION:
Hypothesis:

The use of local anesthetic or vibrating instrument will decrease overall pain experienced by a patient with spasmodic dysphonia undergoing Botox injections.

Aims, purpose, or objectives:

To identify adjuvant methods to improve patient comfort during in-office laryngology procedures. Results demonstrated here should be transferrable to other transcutaneous in-office procedures in laryngology.

Background:

Spasmodic dysphonia is a vocal disorder characterized by uncontrollable voice breaks. Injection of botulinum neurotoxin into the laryngeal muscles is the mainstay of treatment. Patients require repeated treatments due to the temporary effect of botulinum neurotoxin. Laryngeal injections are commonly performed through the skin of the neck and can be associated with pain and discomfort. Local anesthetic administration prior to laryngeal injection is commonly performed in clinical practice, however its efficacy hasn't been evaluated and a third of surveyed otolaryngologists do not administer local anesthesia prior to the laryngeal injection of botulinum neurotoxin. Vibratory anesthesia involves the application of a local vibratory stimulus and has been found to reduce pain during various needle-related procedures. Vibratory anesthesia has not previous been evaluated for laryngeal injections.

This study will utilize the need for spasmodic dysphonia patients to receive repeated injections to incorporate a crossover design where patients receive three consecutive laryngeal injections of botulinum toxin experiencing injection without additional anesthesia, with local anesthesia, and with vibration anesthesia in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

* Spasmodic dysphonia with or without tremor
* Receiving botox as treatment via a transcricothyroid approach

Exclusion Criteria:

- Allergy to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lott, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 32 participants were enrolled to receive all interventions; however, the order the intervention that was received was randomized. All subjects completed all study visits/interventions.
Groups:
- Control, Then Lidocaine, Then Vibrating Wand: At the first injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach without additional anesthesia. At the second injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach following subcutaneous injection of lidocaine (approximately 2 minutes before Botox injection). At the third injection Patients will receive standard of care laryngeal injection of Botox via a transcricothyroid approach while using the vibrating wand.
  Lidocaine: Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
  Vibrating wand: a vibrating instrument held adjacent to the cricothyroid space
- Control, Then Vibrating Wand, Then Lidocaine: At the first injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach without additional anesthesia. At the second injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach while using the vibrating wand. At the third injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach following subcutaneous injection of lidocaine (approximately 2 minutes before Botox injection).
  Vibrating wand: a vibrating instrument held adjacent to the cricothyroid space
  Lidocaine: Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
- Lidocaine, Then Vibrating Wand, Then Control: At the first injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach following subcutaneous injection of lidocaine (approximately 2 minutes before Botox injection). At the second injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach while using the vibrating wand. At the third injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach without additional anesthesia.
  Lidocaine: Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
  Vibrating wand: a vibrating instrument held adjacent to the cricothyroid space
- Lidocaine, Then Control, Then Vibrating Wand: At the first injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach following subcutaneous injection of lidocaine (approximately 2 minutes before Botox injection). At the second injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach without additional anesthesia. At the third injections subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach while using the vibrating wand.
  Lidocaine: Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
  Vibrating wand: a vibrating instrument held adjacent to the cricothyroid space
- Vibrating Wand, Then Control, Then Lidocaine: At the first injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach while using the vibrating wand. At the second injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach without additional anesthesia. At the third injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach following subcutaneous injection of lidocaine (approximately 2 minutes before Botox injection).
  Vibrating wand: a vibrating instrument held adjacent to the cricothyroid space
  Lidocaine: Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
- Vibrating Wand, Then Lidocaine, Then Control: At the first injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach while using the vibrating wand. At the second injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach following subcutaneous injection of lidocaine (approximately 2 minutes before Botox injection). At the third injection subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach without additional anesthesia.
  Vibrating wand: a vibrating instrument held adjacent to the cricothyroid space
  Lidocaine: Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
Period: First Experimental Visit
Arm/Group | Control, Then Lidocaine, Then Vibrating Wand | Control, Then Vibrating Wand, Then Lidocaine | Lidocaine, Then Vibrating Wand, Then Control | Lidocaine, Then Control, Then Vibrating Wand | Vibrating Wand, Then Control, Then Lidocaine | Vibrating Wand, Then Lidocaine, Then Control
Started | 5 | 8 | 6 | 5 | 2 | 6
Completed | 5 | 8 | 6 | 5 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Experimental Visit
Arm/Group | Control, Then Lidocaine, Then Vibrating Wand | Control, Then Vibrating Wand, Then Lidocaine | Lidocaine, Then Vibrating Wand, Then Control | Lidocaine, Then Control, Then Vibrating Wand | Vibrating Wand, Then Control, Then Lidocaine | Vibrating Wand, Then Lidocaine, Then Control
Started | 5 | 8 | 6 | 5 | 2 | 6
Completed | 5 | 8 | 6 | 5 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Experimental Visit
Arm/Group | Control, Then Lidocaine, Then Vibrating Wand | Control, Then Vibrating Wand, Then Lidocaine | Lidocaine, Then Vibrating Wand, Then Control | Lidocaine, Then Control, Then Vibrating Wand | Vibrating Wand, Then Control, Then Lidocaine | Vibrating Wand, Then Lidocaine, Then Control
Started | 5 | 8 | 6 | 5 | 2 | 6
Completed | 5 | 8 | 6 | 5 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total of 32 participants were enrolled to receive all interventions; however, the order the intervention was received was randomized. All 32 subjects completed all study visits/interventions.
Groups:
- Laryngeal Injection of Botox Via a Transcricothyroid Approach: Subjects were randomized at screening to either receive nothing (control), Lidocaine injection prior to their Botox injection or Vibrating Wand held to their skin during the botox injection. Subjects attended three visits of the experiment on three separate days. For the three visits, the subjects received either nothing (control), Lidocaine injection prior to their Botox injection or Vibrating Wand held to their skin during the botox injection, (the order was randomized)
  Lidocaine: Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
  Vibrating wand: a vibrating instrument held adjacent to the cricothyroid space
Arm/Group | Laryngeal Injection of Botox Via a Transcricothyroid Approach
Number analyzed (Participants) | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [61 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Pain Experienced
Description: Measured on a Visual Analogue Scale where 0 = no pain and 10 = worst pain
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Laryngeal Injection of Botox Via a Transcricothyroid Approach
Number analyzed (Participants) | 32
score on a scale
  Control | 2 [1 to 3]
  Lidocaine | 2 [1 to 3.5]
  Vibrating Wand | 2 [1 to 3]

2. Secondary Outcome: Subject Preference
Description: Subjects were asked which technique (Control, Lidocaine or Vibrating wand) they preferred the most
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Laryngeal Injection of Botox Via a Transcricothyroid Approach
Number analyzed (Participants) | 32
Participants
  Control | 6
  Lidocaine | 12
  Vibrating Wand | 14

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for all subjects for the first experimental visit, second experimental visit and third experimental visit to end of study for a total of approximately 6 months.
Groups:
- Control: Subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach without additional anesthesia at either the first, second, or third experimental visit
- Lidocaine: Subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach followed by subcutaneous injection of lidocaine (approximately 2 minutes before Botox injection) at either the first, second, or third experimental visit
  Lidocaine: Subcutaneous injection 0.5cc 2% in 1:100,000 epinephrine
- Vibrating Wand: Subjects received standard of care laryngeal injection of Botox via a transcricothyroid approach while using the vibrating wand at either the first, second, or third experimental visit
  Vibrating wand: a vibrating instrument held adjacent to the cricothyroid space
Arm/Group | Control | Lidocaine | Vibrating Wand
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT04648891/Prot_SAP_000.pdf